CLINICAL TRIAL: NCT04891510
Title: A Comparative Analysis of REVOLVE, LipoGrafter, and Viality in Autologous Fat Grafting During Breast Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-10022850
Record Dates: First submitted 2021-05-17; First posted 2021-05-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mastectomy; Mammaplasty; Breast Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- REVOLVE Advanced Adipose System (Active Comparator): Participants will receive the REVOLVE Advanced Adipose System technique during breast reconstruction.
  Interventions: Device: REVOLVE Advanced Adipose System
- LipoGrafter (Active Comparator): Participants will receive the LipoGrafter technique during breast reconstruction.
  Interventions: Device: LipoGrafter
- Viality (Active Comparator): Participants will receive the Viality technique during breast reconstruction.
  Interventions: Procedure: Viality

INTERVENTIONS:
Device: REVOLVE Advanced Adipose System — The REVOLVE system is an all-in-one fat processing device that harvests, filters, actively washes, and removes strands from lipoaspirate and allows for reinjection without any additional manipulation (REVOLVE 2020).
  Arms: REVOLVE Advanced Adipose System
Device: LipoGrafter — The LipoGrafter system is designed to be a start-to-finish closed system with minimal processing of the lipoaspirate, minimizing the risk of contamination and fat cell damage (LipoGrafter 2020).
  Arms: LipoGrafter
Procedure: Viality — The Viality system uses the AuraClens solution that acts as a surfactant to bring impurities like blood, free oil, and cellular debris into solution, where they can be flushed out through suction.
  Arms: Viality

SUMMARY:
The purpose of this study is to learn whether there is a superior fat processing method in terms of graft retention in breast reconstruction after mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Documented history of previous breast surgery (either complete or partial mastectomy);
* Available harvest sites for fat grafting as documented by plastic surgeon;
* BMI > 20;
* Anticipated harvested fat volume > 50cc;
* Competency and willingness to provide consent

Exclusion Criteria:

* Suspected or known to be pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in efficacy of fat grafting technique, as measured by 3D volumetric scanning at the surgical site | Baseline, 90 day follow-up
  3D volumetric scanning assesses the fat graft retention defined as the ratio of fat remaining at the surgical site at 90 day follow-up to that at pre-operative baseline.
Change in patient satisfaction of fat grafting technique, as measured by the BREAST-Q questionnaire | Baseline, 90 day follow-up
  The BREAST-Q questionnaire is used for measuring pre- and postoperative psychosocial, physical, and sexual well-being, satisfaction with breasts, experience of care, and satisfaction with outcome. Scores range on a 0-100 scale, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Number of palpable masses from the fat grafting technique, as measured by a physical exam. | 90 day follow-up
  The physical exam will provide the number of palpable masses at the surgical site.
Number of lesions of probable fat necrosis from the fat grafting technique, as measured by a physical exam | 90 day follow-up
  The physical exam will provide the number of lesions of probable fat necrosis at the surgical site
Presence of infection from the fat grafting technique, as measured by a physical exam | 90 day follow-up
  The physical exam will show if there is infection present at the surgical site. This is a binary "yes/no" item.
Presence seroma from the fat grafting technique, as measured by a physical exam | 90 day follow-up
  The physical exam will show if there is seroma present at the surgical site. This is a binary "yes/no" item.
Assessment of wound healing from the fat grafting technique, as measured by a physical exam | 90 day follow-up
  The physical exam will show if wound healing is normal or delayed at the surgical site. This is a binary "normal/delayed" item.

CONTACTS AND LOCATIONS:
Overall Officials: David Otterburn, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian - Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No